CLINICAL TRIAL: NCT02537990
Title: MDS-CAN: A Prospective National MDS Clinical Database and Local Tissue Bank
Acronym: MDS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: Tom Baker Cancer Centre (Other); CancerCare Manitoba (Other); The Ottawa Hospital (Other); Princess Margaret Hospital, Canada (Other); Jewish General Hospital (Other); Health Sciences Centre, Winnipeg, Manitoba (Other); British Columbia Cancer Agency (Other); Providence Health & Services (Other); Vancouver Coastal Health (Other Government); Juravinski Cancer Center (Other); Réseau de Santé Vitalité Health Network (Other); Royal Victoria Hospital, Canada (Other); Capital Health, Canada (Other); Saskatoon City Hospital (Other)
Responsible Party: Principal Investigator, Dr. Rena Buckstein, Head Hematology Site Group, Sunnybrook Health Sciences Centre
Other Study IDs: MDS Database
Record Dates: First submitted 2015-08-19; First posted 2015-09-02 (Estimated); Last update posted 2016-11-16 (Estimated); Status verified 2016-11

CONDITIONS: Myelodysplastic Syndrome (MDS)
MeSH Terms: conditions — Myelodysplastic Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Years
Biospecimen Retention: Samples With DNA — Specimens of bone marrow will be collected by aspiration when bone marrows are done for clinical purposes only. BM Plasma will be stored in aliquots, Mononuclear cells (MCs) will be isolated by density gradient centrifugation of buffy coat cells. The remainder of MC collected in this way will be used for immediate extraction of DNA by standard techniques.
Oversight: Data Monitoring Committee: No

SUMMARY:
The purposes of this study are: 1. To identify and quantify the health utilities and quality of life experienced by patients who have been diagnosed with MDS and what are their predictors. 2. Measure the effects of patient related factors like frailty and comorbidity on quality of life and overall survival or toxicity to therapy. 3. Assess how quality of life changes over time and what are its predictors. This will be valuable information that may guide therapy, transfusion practices, etc., as MDS is a chronic, incurable disease that is often progressive.

DETAILED DESCRIPTION:
o Participants will be seen and assessed for the study every 6 (+/-1) months. Follow-up for routine clinical care will be dictated by the physician. Clinical information relevant to the MDS diagnosis is entered such as IPSS, IPSS-R, treatments received and responses. Transfusion dependence is recorded. Relevant laboratories such as ferritin, LDH, CBC etc are entered q 6 months. Hospitalizations, bleeding and infections are recorded.

Dates and causes of death are documented Dates of leukaemia transformation are documented. Patients undergoing allogeneic stem cell transplant are documented with date of transplant.

QOL is assessed every 6 months:

QOL instruments are QLQ-C30, QUALMS, EQ-5D and global fatigue scale

Disability, frailty, comorbidity and physical performance is recorded on a yearly basis Disability scale is the Lawton Brody SIADL scale Frailty is measured using the Rockwood clinical frailty scale The comorbidity elements necessary to calculate the Charlson comorbidity scale and the MDS-CI of Della Porta et al. are recorded Physical performance tests are grip strength, 10x stand sit test and the 4 meter walk test

Investigators will continue to enroll new patients throughout this study period of 6 years, but the plan (funding permitting) is to continue this registry indefinitely, with later questions to be addressed.

* Monitoring and auditing data are completed every quarter by a dedicated national registry project manager.
* Monthly data checks are completed to compare data entered into the registry against predefined rules for range or consistency with other data fields in the registry.
* Standard Operating Procedures to address registry operations and analysis activities, such as patient recruitment and data collection has been created and posted electronically in the database for all sites.
* Plan of 25% drop off from death has been assumed due to conversion to AML or non leukemia death and 5% from lost of follow up loss to follow up. This is with the purpose to address situations where variables are reported as missing, unavailable, "non-reported," uninterpreted, or considered missing because of data inconsistency or out-of-range.
* Participant's results will be summarized descriptively as a whole and by province. KM survival curves will be generated and compared using the log-rank test. Univariate and multivariate cox proportional hazard nodel of overall survival will be performed to detect significant association with baseline covariates and time-dependent covariates such as frailty, comorbidity and QOL scores using Statistical Analysis Software (SAS) PHREG procedure.

ELIGIBILITY:
Inclusion Criteria:

* New diagnosis of a Myelodysplastic syndrome
* New diagnosis of CMML-1/CMML-2 and MDS/MPN
* New diagnosis of low blast AML (blasts 20-30%) as defined by the WHO classification (Vardiman, 2002)
* Greater than 18 years of age at the time of diagnosis
* Able to read, write and speak English or French (non-English or French speaking patients may participate if appropriate translation is used)
* Able to consent.

Exclusion Criteria:

* Patients whose diagnostic bone marrow exceed 2 years prior signing consent
* Subjects with AML and bone marrow blast of 31% or more at the time of signing consent
* Prior allogenic cell transplant

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary care clinic, referrals from community physicians.
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2005-08; Primary Completion 2020-02 (Estimated); Study Completion 2020-02 (Estimated)

PRIMARY OUTCOMES:
quality of life | every 6 months up to 6 years

CONTACTS AND LOCATIONS:
Overall Officials: Rena Buckstein, MD FRCPC, Study Director — Sunnybrook Health Science Centre
Locations (1):
- Odette Cancer Center, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data can be available to other researchers for their own patients from that center but not other centers. Collective anonymized data of all registry patients is available to them however.

REFERENCES:
- [Derived] Buckstein R, Chodirker L, Mozessohn L, Yee KWL, Geddes M, Zhu N, Shamy A, Leitch HA, Christou G, Banerji V, Brian L, Khalaf D, St-Hilaire E, Finn N, Nevill T, Keating MM, Storring J, Delage R, Parmentier A, Thambipillai A, Siddiqui M, Westcott C, Cameron C, Mamedov A, Spin P, Tang D. A natural history of lower-risk myelodysplastic syndromes with ring sideroblasts: an analysis of the MDS-CAN registry. Leuk Lymphoma. 2022 Dec;63(13):3165-3174. doi: 10.1080/10428194.2022.2109154. Epub 2022 Sep 12. PMID 36095125
- [Derived] Buckstein R, Wells RA, Zhu N, Leitch HA, Nevill TJ, Yee KW, Leber B, Sabloff M, St Hilaire E, Kumar R, Geddes M, Shamy A, Storring J, Kew A, Elemary M, Levitt M, Lenis M, Mamedov A, Zhang L, Rockwood K, Alibhai SM. Patient-related factors independently impact overall survival in patients with myelodysplastic syndromes: an MDS-CAN prospective study. Br J Haematol. 2016 Jul;174(1):88-101. doi: 10.1111/bjh.14033. Epub 2016 Mar 15. PMID 26991631